CLINICAL TRIAL: NCT05330754
Title: Effect Of Daily Caffeine Intake On Perioperative Analgesic Consumption And Recovery Time In Patients Undergoing Laparoscopic Surgeries.
Brief Title: Caffeine Intake Inrelation to Perioperative Analgesic Consumption
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor of Anesthesia, Ain Shams University
Other Study IDs: R 67/ 2022
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Analgesia; Caffeine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: No caffeine intake
  Interventions: Dietary Supplement: Caffeine intake in mg
- Safe level Group: Caffeine daily intake ≤200 mg/day
  Interventions: Dietary Supplement: Caffeine intake in mg
- Unsafe level group:: Caffeine daily intake >200 mg/day
  Interventions: Dietary Supplement: Caffeine intake in mg

INTERVENTIONS:
Dietary Supplement: Caffeine intake in mg — Preanesthetic check-up was done. Average daily caffeine consumption in mg was calculated according to "caffeine content in consumed drinks" as estimated by "Food Data Central".

SUMMARY:
Caffeine is the most widely consumed psychoactive drug in the world. Natural sources of caffeine include coffee, tea, and chocolate. Synthetic caffeine is also added to products to promote arousal, alertness, energy, and elevated mood.

We designed this prospective observational study to determine if caffeine consumption would influence intraoperative analgesic consumption

DETAILED DESCRIPTION:
Caffeine is a well-known natural compound present in various plant products. Caffeine is an integral component of several daily drinks, including tea, coffee, soft drinks, and energy drinks [1]. (e consumption habits of these caffeinated drinks have facilitated the wide distribution of and dependence on caffeine. For instance, 89% of the US adult population has an average caffeine intake of 200 mg/day [2]. Among the multiple effects and side effects, caffeine also has an analgesic action and is used to reduce pain in several pharmaceutical forms as an adjuvant [1]. Several studies have reported a role for caffeine in controlling pain and suggested that caffeine may block the central processing of pain signals in the brain and enhance the body's natural pain resistance pathways [3]. In addition, Overstreet et al. found that habitual caffeine consumption diminishes pain sensitivity in a laboratory setting [4]

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective laparoscopic surgery

Exclusion Criteria:

* Patients converted to an open surgery, postoperative complications that increased postoperative pain, and those with psychological or nervous system diseases were also excluded. Liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 - 65 years old, physical status American Society of Anesthesiology (ASA) I&II, body weight from 70-80 kg,
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
total intraoperative fentanyl consumption in microgram | 2 hours
  Amount of total intraoperative fentanyl consumption in microgram

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request